CLINICAL TRIAL: NCT04222127
Title: EUS-Guided Cyanoacrylate Injection Versus Standard Endoscopic Technique in the Obturation of High Risk Gastric Varices
Brief Title: EUS-guided Obturation of High Risk Gastric Varices Versus Standard Endoscopic Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MD.19.03.157
Record Dates: First submitted 2019-10-05; First posted 2020-01-09 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Gastric Varix
Keywords: Gastric Varices; EUS; Cyanoacrylate
MeSH Terms: conditions — Esophageal and Gastric Varices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EUS-guided injection of CYA of GVs (Experimental): EUS-guided injection of CYA will be done at entrance of of the varix or the perforator veins when identifiable using a mixture (1:1) of 2-octyl-cyanoacrylate & lipidol using 19G EUS-FNA needle
  Interventions: Other: EUS guided injection of gastric varices by CYA
- Direct endoscopic injection of CYA of GVs (Experimental): Direct endoscopic injection of CYA of the gastric varix using standard endoscopy
  Interventions: Other: Direct endoscopic injection of gastric varices by CYA

INTERVENTIONS:
Other: EUS guided injection of gastric varices by CYA — EUS-guided injection of CYA will be done at entrance of of the varix or the perforator veins when identifiable using a mixture (1:1) of 2-octyl-cyanoacrylate & lipidol using 19G EUS-FNA needle
  Arms: EUS-guided injection of CYA of GVs
Other: Direct endoscopic injection of gastric varices by CYA — Direct endoscopic injection of gastric varix by CYA
  Arms: Direct endoscopic injection of CYA of GVs

SUMMARY:
Gastric varices occur in patients with portal hypertension, mostly secondary to liver cirrhosis. Although they bleed less frequently than oesophageal varices, gastric variceal bleeding tends to be more severe with reported higher mortality.

Endoscopic variceal obliteration (EVO) by direct endoscopic injection (DEI) using tissue adhesives like glue, CYA or histoacryl demonstrated higher hemostasis and lower bleeding rates compared to band ligation or sclerotherapy. Nevertheless, CYA treatment is known to be associated with significant adverse events like para-variceal injection, hemorrhage from post injection ulcer, needle sticking in the varix, intra-peritoneal injection leading to peritonitis and adherence of the glue to the endoscope, fever, embolization into the renal vein, IVC, pulmonary or systemic vessels.

Endoscopic ultrasound (EUS) offers unique access to abdominal arterial and venous vasculature. This has had the most clinical impact on the treatment of gastroesophageal varices, where EUS may play a role both in the management and can deliver therapy in the form of glue injection, endovascular coil placement or a combination of the two. EUS enables an assessment using Doppler to confirm vessel obliteration after treatment. However, targeting the perforating feeder vessel rather than the varix lumen itself may theoretically minimize the amount of CYA needed to achieve obliteration of GVs and thereby reduce the risk of embolization.

DETAILED DESCRIPTION:
This is a single-centre, pilot randomized trial study that includes 42 patients with gastric varices that will be classified according to the Sarin and Kumar classification into GOV II or IGV I with recently bleeding GV & high-risk GV (defined by Baveno VI consensus for primary prophylaxis).

Eligible patients will be randomized in 2 groups using computer-generated random number sequences using excel software in concealed envelopes with block randomization design. Group I will undergo EUS-guided CYA injection at entrance of perforator veins. Group II will undergo DEI of CYA.

Each patient will be subjected to :

* Written informed consent will be obtained from each patient, including a discussion on the procedure.
* Clinical assessment including history taking and physical examination
* Routine laboratory investigations including complete blood picture and serum creatinine.
* Liver function profile (serum bilirubin, AST, ALT , albumin and prothrombin time).
* The severity of underlying disease will be assessed by the Child-Turcotte-Pugh score (CTP) based on serum albumin, bilirubin, prothrombin time, the presence of ascites and encephalopathy.
* All procedures will be performed under deep sedation or general anesthesia in the left lateral position.
* Intravenous antibiotics will be administered to all patients prior to the endoscopic procedure to minimize the risk of secondary bacterial infection. Oral or intravenous antibiotics will be continued for at least 3 days following variceal injection.

  * Endoscopic procedure and technique:
* Standard diagnostic upper endoscopy will be performed in order to classify the varices according to the classification of Sarin and Kumar. Only high risk GOV II and IGV I varices (>10 mm) will be included.
* EUS examination will be done in all patients with a Pentax linear Echoendoscope EG3870UTK (PENTAX medical, Tokyo, Japan) attached to a Hitachi Avius ultrasound system (Hitachi Medical Systems, Tokyo, Japan). All EUS examinations will be done by two endosonographers. The echoendoscope will be positioned in the distal esophagus at the level of the cardia to visualize the gastric fundus and intramural varices.
* EUS will be used to display the vascular anatomy, in particular the feeding vein. GVs will be classified endosonographically according to Boustière et al which considered size of GVs and gastric wall abnormalities :

  1: Size of GVs:
* Grade 0 (none)
* Grade 1 (small or non-confluent varies < 5 mm)
* Grade 2 (large or confluent varices ≥ 5 mm) 2: Abnormalities of gastric wall:

  1. Grade 0 (none)
  2. Grade 1 (thickening and brilliance of the third hyperechogenic layer with or without fine internal anechogenic structures).
  3. Grade 2 (visible vessels in the third layer which deform the entire wall, with penetrating varices).
* EUS-guided injection of CYA will be done at entrance of of the varix or the perforator veins when identifiable using a mixture (1:1) of 2-octyl-cyanoacrylate & lipidol using 19G EUS-FNA needle in Group I, or DEI of CYA in Group II.

  * Follow-up after endoscopy:

After the procedure, patients will be observed for 2 hours in the recovery room before being discharged. Endoscopic examination and Doppler EUS will be repeated in all patients at 3, and 6 months post-procedure (or sooner with recurrent bleeding) to confirm eradication. Hemostasis, early post treatment bleeding and late post treatment bleeding will be recorded according to Baveno VI concensus.

GVs will be considered obliterated by direct endoscopy when not visible and/or hardened to catheter palpation. Obliteration by Doppler EUS will be considered by visualization of clot and absence of Doppler flow within the gastric wall. Repeat injection will be performed in the absence of obliteration. Direct endoscopic and Doppler EUS examinations will be repeated again at 3, and 6 months after each injection.

ELIGIBILITY:
Inclusion Criteria:

* High risk GOV II and IGV I varices (>10 mm) on initial standard diagnostic upper endoscopy
* Recent bleeding and primary prophylaxis
* Patients who are unable or unwilling to undergo alternative therapies for GV [such as transjugular intrahepatic portosystemic shunts (TIPS) or surgery], or prior TIPS had failed.

Exclusion Criteria:

* Inability to give informed consent for the procedure.
* Concurrent hepatorenal syndrome and/or multiorgan failure.
* Presence of HCC &/or portal vein thrombosis.
* Previous endoscopic treatment for GVs.
* Platelet count less than 50,000/ml or International Normalized Rate (INR) >2
* Esophageal stricture
* Previous esophageal or gastric surgery.
* Pregnancy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events & oblitration rate | 6 months
  measure the technical success rate defined as complete variceal obliteration and complications rate including bleeding, pulmonary embolism (PE), ulcers, fever, paravariceal injection & rebleeding.

SECONDARY OUTCOMES:
Amount of glue used | 6 months
  amount of cyanoacrylate used to complete obliteration in ml.
Number of sessions | 6 months
  calculate the number of sessions needed to achieve oblitration of gastric varices

CONTACTS AND LOCATIONS:
Overall Officials: Fady S Karam, Master, Principal Investigator — Mansoura University; Ahmed Y Altonbary, MD, Study Director — Mansoura University; Hazim H Almenshawy, Professor, Study Director — Mansoura University; Ayman A Aldosoky, Professor, Study Director — Mansoura University; Seham M Seif, Professor, Study Chair — Mansoura University
Locations (1):
- Specialized Medical hospital, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Romero-Castro R, Pellicer-Bautista FJ, Jimenez-Saenz M, Marcos-Sanchez F, Caunedo-Alvarez A, Ortiz-Moyano C, Gomez-Parra M, Herrerias-Gutierrez JM. EUS-guided injection of cyanoacrylate in perforating feeding veins in gastric varices: results in 5 cases. Gastrointest Endosc. 2007 Aug;66(2):402-7. doi: 10.1016/j.gie.2007.03.008. PMID 17643723
- [Background] Wang AJ, Li BM, Zheng XL, Shu X, Zhu X. Utility of endoscopic ultrasound in the diagnosis and management of esophagogastric varices. Endosc Ultrasound. 2016 Jul-Aug;5(4):218-24. doi: 10.4103/2303-9027.187840. PMID 27503152

DOCUMENTS (1):
  • Study Protocol (2019-01-01): https://cdn.clinicaltrials.gov/large-docs/27/NCT04222127/Prot_000.pdf